CLINICAL TRIAL: NCT03461393
Title: The Effects of Regular Eye-training With a Mobile Device on Adult Patients With AMD
Acronym: ETAMD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Applied Sciences Upper Austria (Other)
Collaborators: Krankenhaus der Barmherzigen Schwestern Ried (Other)
Responsible Party: Principal Investigator, Thomas Haslwanter, Prof.(FH) Dr., University of Applied Sciences Upper Austria
Other Study IDs: Uasua
Record Dates: First submitted 2018-03-05; First posted 2018-03-12 (Actual); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: AMD
Keywords: AMD; Mobile Device; Training

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intervention Group: Repetitive Training with Medical-Eye-Trainer (MET)
  Interventions: Device: Medical-Eye-Trainer (MET)

INTERVENTIONS:
Device: Medical-Eye-Trainer (MET) — In order to provide a high contrast, dynamic visual stimulus to the patients, we developed an app that allowed the patients to regularly train with this stimulus. The app runs on Android (version 4.2 or later). The display of the screen is divided into 4 rows. In each row, a pattern of black and white squares is moving in one direction. The directions in subsequent rows are opposite to each other. Through the movement in the opposite direction a changing pattern is achieved in vertical and horizontal extension, the pattern alternates between continuous beams and a checkered pattern. The speed of the display on the monitor is 2 cm per second. In a comfortable viewing distance (ca. 40 cm), this leads to an angular velocity of approximately 3°/sec.

SUMMARY:
Data collection and observation of changes within AMD patients performing visual training on mobile devices

DETAILED DESCRIPTION:
In the presented study a training-therapy in patients with dry AMD war evaluated. The main focus was on remote visibility and thus better handling of daily activities.

Therapy with high-contrast administration is used for amblyopia in childhood. Furthermore, simulation therapy is used in hemianopsia in the adult age, in which case the lesion is usually not located in the eye.

This stimulating therapy for children and adult patients led to the hypothesis that this treatment could also improve AMD's situation. The entire visual procedure also shows the possibility of change even in adult patients.

The presented study investigates if regular training with a device that provides a moving grating-stimulus, the "Medical Eye Trainer" (MET), can improve the subjective perception of visual performance during typical activities of daily living. The aims of the study were not to show improvement of reading vision nor to show changes in the retinal structure.

ELIGIBILITY:
Inclusion Criteria:

* All eyes had been affected by dry AMD for 3.5 years or more

Exclusion Criteria:

None

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In the study, 11 patients were included. In five of those, both eyes were affected by AMD; in the six other patients, only one eye was affected. The age of the patients was 72 ± 14.7 years (mean ± standard deviation, range 44 - 86 years). Eight eyes had received a lutein therapy for more than 2 years, according to the Age-Related Eye Diseases Study (AREDS) study. In two eyes an anti-VEGF (vascular endothelial growth factor ) therapy had been performed before (3.5 and 4 years ago, respecitvely); and in one eye a photodynamic therapy (PDT) had been performed 9 years ago. All eyes had been affected by dry AMD for 3.5 years or more. The visual acuity had been unchanged for at least a year in all patients. None of the patients reported any previous occurrence of epilepsy.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Estimated)
Dates: Start 2018-04-01 (Estimated); Primary Completion 2018-04-30 (Estimated); Study Completion 2018-05-15 (Estimated)

PRIMARY OUTCOMES:
Visual Acuity | Baseline - 3 months
  6 meter - Decimal

SECONDARY OUTCOMES:
Subjective Satisfaction | Baseline - 3 months
  better - no Change - worse

CONTACTS AND LOCATIONS:
Locations (1):
- Krankenhaus der Barmherzigen Schwestern Ried, Ried im Innkreis, Upper Austria, Austria

IPD SHARING:
Plan to Share IPD: No